CLINICAL TRIAL: NCT00213694
Title: Efficacy of Docetaxel (J 15) and Celecoxib in Metastatic Prostate Cancer
Brief Title: PROSTACOX : Metastatic Prostate Chemotherapy
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Other Study IDs: 2003/052/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Celecoxib

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: docetaxel and celecoxib

SUMMARY:
Clinical response to chemotherapy. Biological parameter (PSA) and RECIST evaluation. Association of Docetaxel (J 15) and Celecoxib.

DETAILED DESCRIPTION:
Association Docetaxel (J 15) and celecoxib Patient survival Biological parameter : PSA Clinical status RECIST evaluation

ELIGIBILITY:
Inclusion Criteria:

* metastatic prostate cancer
* ASCO progression criteria

Exclusion Criteria:

* other prostate chemotherapy

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52
Dates: Start 2003-11; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Christian PFISTER, MD, PhD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Charles Nicolle, University Hospital, Rouen, France